CLINICAL TRIAL: NCT07111000
Title: Evaluating the Efficacy of Epley Maneuver in the Treatment of Benign Paroxysmal Positional Vertigo in the Emergency Department: A Randomized Controlled Trial.
Brief Title: Testing the Epley Maneuver for Treating Dizziness in the Emergency Department: A Randomized Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Eveline Hitti, Professor of Clinical Specialty, American University of Beirut Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2023-0184
Record Dates: First submitted 2025-08-06; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-12

CONDITIONS: Benign Paroxysmal Positional Vertigo (BPPV)
Keywords: Benign Paroxysmal Positional Vertigo (BPPV), vertigo, Epley maneuver, Dix-Hallpike Test (DHT)
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epley Maneuver (Experimental): The patient's head is turned 45 degrees towards the side that caused the most nystagmus or reproduced their initial symptoms. The patient is then laid down with their head hanging over the edge of the bed. After that, the head will be rotated 90 degrees in the opposite direction, with the head remaining in a dependent position. The patient is then asked to roll onto their side with their head facing downward. They are then brought back to a sitting position and the head is moved forward 45 degrees. Each position is held until the vertigo and/or nystagmus subsides or for at least 30 seconds
  Interventions: Procedure: Epley Maneuver
- Sham Maneuver (Sham Comparator)
  Interventions: Procedure: Sham maneuver

INTERVENTIONS:
Procedure: Epley Maneuver — The patient's head is turned 45 degrees towards the side that caused the most nystagmus or reproduced their initial symptoms. The patient is then laid down with their head hanging over the edge of the bed. After that, the head will be rotated 90 degrees in the opposite direction, with the head remaining in a dependent position. The patient is then asked to roll onto their side with their head facing downward. They are then brought back to a sitting position and the head is moved forward 45 degrees. Each position is held until the vertigo and/or nystagmus subsides or for at least 30 seconds
  Arms: Epley Maneuver
Procedure: Sham maneuver — This control maneuver will involve coordinated movements of the hands and legs, while excluding any head movement. Patients will be at first in a sitting position with both feet on the ground and both hands placed on the thighs and then they will be asked to lift both hands off the thighs, keeping the arms extended. They will then be asked to return to their initial upright sitting position. Patients will then raise their right foot off the ground while keeping the left one planted on the ground. It will be an alternating movement between lifting the right and left feet while maintaining a smooth and well- controlled rhythm for 90 seconds.
  Arms: Sham Maneuver

SUMMARY:
The goal of this randomized controlled trial is to evaluate the efficacy of the Epley maneuver versus a sham maneuver in treating patients presenting to the emergency department (ED) with BPPV. The main questions that the study aims to answer are:

* What is the mean difference in Dizziness Handicap Inventory (DHI) scores between patients receiving the Epley maneuver and those receiving the sham maneuver 3 days after enrollment?
* What is the immediate response (using a 0-10-point Likert scale) of patients in each arm of the study?
* What is the proportion of patients who, despite agreeing to participate, were unable to complete the full Epley maneuver due to symptom severity?

Researchers will compare the Epley maneuver arm to the sham maneuver arm to see if the Epley maneuver is more effective in reducing BPPV symptoms.

Participants will:

* Undergo either the Epley maneuver or a sham maneuver.
* Complete the Dizziness Handicap Inventory (DHI) questionnaire at baseline and 3 days post-discharge.
* Patients with insufficient improvement in the sham maneuver group will receive a rescue Epley maneuver.
* Have their vertigo severity assessed using a 0-10 point Likert scale at baseline, immediately and post-maneuver.

ELIGIBILITY:
Patients presenting to the ED with symptoms of BPPV (single or recurrent episodes of vertigo lasting up to 2 minutes) and a positive DHT (episode of vertigo associated with torsional upbeating nystagmus) indicating a posterior semicircular canal BPPV.

Patients who are able to understand and provide a signed informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Epley | 3 days
  The study will compare the average Dizziness Handicap Inventory score change from baseline to day 3 between the Epley maneuver group and the sham maneuver group.

SECONDARY OUTCOMES:
Immediate response of patients | 15-30 minutes after intervention
  The severity of vertigo will be evaluated using both a 0 to 10-point Likert scale before and after applying the Epley/Sham maneuver.
Rate of bounce-back to the ED | 3 days
  Calculate the proportion of patients in each arm of the study who return to the ED.
Proportion of patients unable to undergo the full Epley maneuver | 15 minutes
  The percentage of patients who agreed to participate but could not complete the Epley maneuver due to the severity of their symptoms.